CLINICAL TRIAL: NCT06923293
Title: Individualizing Powered Orthotic Intervention for Improved Gait Outcomes Using ML-enabled Methods
Brief Title: Improving Walking After a Lower Limb Injury Using a Custom Motorized Orthosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: Stevens Institute of Technology (Other)
Responsible Party: Principal Investigator, Karen J. Nolan, PhD, Associate DIrector, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-1182-22
Record Dates: First submitted 2025-04-02; First posted 2025-04-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Lower Limb Injury
MeSH Terms: conditions — Leg Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Adults with lower limb injury (Experimental): All enrolled subjects will be asked to complete the intervention.
  Interventions: Device: Utilization of motorized orthosis

INTERVENTIONS:
Device: Utilization of motorized orthosis — While part of this study, participants will be fitted for the motorized orthosis and will complete walking tests with and without the AFO.

SUMMARY:
The purpose of this research study is to assess the ease, convenience, and efficacy of walking when using a motor powered ankle foot orthosis (AFO) brace, in adults who have had a lower limb injury.

DETAILED DESCRIPTION:
The long-term goal of this project is to improve the outcomes of robot-assisted exercise interventions for patients with reconstructed lower limb following high-energy lower extremity traumas using novel machine learning methods to enable individualized ankle foot orthosis (AFO) designs and self-adaptive AFO assistance.

The main hypothesis predicts greater comfort and lower pain levels when using the new AFO as well as improvements in gait mechanics, which will outperform those induced by patients' daily-use AFOs. The main goal is this adaptive assistance will encourage the wearer's active engagement in RAGT thereby promoting patient self-efficacy/satisfaction and leading to improvements in ambulation after a 6-week rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Have a lower limb injury greater than a year ago.
* Be 18-80 years old.
* Be able to stand for 30 minutes.
* Have enough range of motion in my ankle to comfortably wear the AFO.
* Be able to follow directions and commands.
* Be willing and able to give informed consent.
* Be able and willing to comply with study procedures, verbal instructions, and follow-up requirements.

Exclusion Criteria:

* Have any joint or muscle tightness that would limit my movement while walking with the AFO.
* Have any medical issue that prevents me from supporting my weight and walking (e.g. orthopedic injuries, pain, severe spasticity).
* Have any medical issues that affect my unaffected side.
* Have skin issues that would prevent wearing the device.
* Have a pre-existing condition that caused exercise intolerance. (Documented uncontrolled hypertension, coronary artery disease, abnormal heart rate or rhythm, or congestive heart failure).
* Have been hospitalized for heart attack, heart surgery or acute heart failure within 3 months of enrollment in study.
* Have nervous system issues that affect my movement (for example Parkinson's disease, multiple sclerosis).
* Have additional orthopedic issues that interfere with my walking or limit my range of motion in my legs.
* Have any other medical conditions that my doctor or physical therapist feels would affect my ability to use the device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
10MWT (Aim 1) | Measured before and after 6 week intervention to assess change from baseline.
  10 meter walk test to evaluate walking speed after lower limb injury and in response to the intervention. Walking evaluated without versus with the motorized orthosis.
TUG (Aim 1) | Measured before and after 6 week intervention to assess change from baseline.
  Timed up and go (TUG) test to measure functional balance and walking ability after lower limb injury and in response to the intervention. Walking evaluated without versus with the motorized orthosis.
6MWT (Aim 1) | Measured before and after 6 week intervention to assess change from baseline.
  6 minute walking test to evaluate endurance after lower limb injury and in response to the intervention. Walking evaluated without versus with the motorized orthosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided